CLINICAL TRIAL: NCT06233318
Title: Efficacy of Bilateral Pecto-Intercostal Fascial Plane Block on Postoperative Pain in Adult Patients Undergoing Open Heart Surgery: a Randomized, Double-blind, Controlled Trial
Brief Title: Sternotomy PIFB Block in Open Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Erica Stein, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023H0076
Record Dates: First submitted 2024-01-12; First posted 2024-01-31 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Autonomic Nerve Block
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized, placebo-controlled, double-blinded trial in patients undergoing open-heart surgery at Richard M. Ross Hospital - The Ohio State University Medical Center. All study procedures will be done in accordance with institutional and ORRP-IRB guidelines.
Who Masked: Participant, Outcomes Assessor
Masking Description: PIFB will be administered to the patient after anesthesia induction and before surgical incision according to the randomization regimen. The unblinded researcher will randomize and inform to the unblinded anesthesia care provider who will perform the PIFB procedure. The rest of clinicians, research personnel and patients will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pecto-intercostal fascial block (Active Comparator): Pecto-intercostal Fascial Block with 20 ml of 0.35% ropivacaine injected to each side under ultrasound visualization.
  Interventions: Procedure: Pecto-intercostal Fascial Block with 20 ml of 0.35% ropivacaine
- Placebo (Placebo Comparator): Pecto-intercostal Fascial Block with 20ml of normal saline injected to each side under ultrasound visualization.
  Interventions: Procedure: Pecto-intercostal Fascial Block with normal saline

INTERVENTIONS:
Procedure: Pecto-intercostal Fascial Block with 20 ml of 0.35% ropivacaine — The US probe will be placed at sagittal plane, 2 cm lateral to the midline of the sternum to identify the second to the fifth costal cartilage from the ribs. Consequently, the US probe will be positioned in the space between the fourth and fifth costal cartilages at the sternum. After identifying the fascial planes of the chest wall, the pectoralis major muscle (PMM), the external intercostal muscle (EIM), the costal cartilage, the pleura, and the lungs. A sterile 22G blunt Stimuplex, 50 mm needle (B. Braun, Bethlehem, Pa) will be advanced and placed under the PMM and above the EIM. Following negative aspiration, PN solution with investigational product according to group randomization/allocation will be injected at each side in 5 mL aliquots ensuring appropriate spread of the PN solution. The separation of the fascial plane and the spread of the drug will be observed on the ultrasound image in real time.
  Arms: Pecto-intercostal fascial block
Procedure: Pecto-intercostal Fascial Block with normal saline — The US probe will be placed at sagittal plane, 2 cm lateral to the midline of the sternum to identify the second to the fifth costal cartilage from the ribs. Consequently, the US probe will be positioned in the space between the fourth and fifth costal cartilages at the sternum. After identifying the fascial planes of the chest wall, the pectoralis major muscle (PMM), the external intercostal muscle (EIM), the costal cartilage, the pleura, and the lungs. A sterile 22G blunt Stimuplex, 50 mm needle (B. Braun, Bethlehem, Pa) will be advanced and placed under the PMM and above the EIM. Following negative aspiration, PN solution with investigational product according to group randomization/allocation will be injected at each side in 5 mL aliquots ensuring appropriate spread of the PN solution. The separation of the fascial plane and the spread of the drug will be observed on the ultrasound image in real time.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if the use of a bilateral nerve block with a local anesthetic (ropivacaine), as part of a standard of care pain control regimen (called multimodal analgesia [MMA]), has a favorable effect on our institutional MMA pain regimen. Subjects will go through the following study procedures: review of medical history and medications subjects have taken within a month prior to surgery. Subjects will be randomly assigned to one of the two study groups (1:1) to receive either, an ultrasound-guided bilateral nerve block (called "Pecto-Intercostal Fascial Block [PIFB]") with ropivacaine or saline 0.9 solution, in addition to our institutional MMA regimen. A baseline line pain and nausea scores will be recorded before surgery. The block will be performed right after general anesthesia induction. The details about the surgery will be collected. Pain assessments, nausea and vomiting scores will be registered at 12, 24 and 48 hours after surgery as well. Lastly, a follow up phone call will be made by the research team to conduct a pain-detect questionnaire at 30, 60 and 90 days after surgery.

DETAILED DESCRIPTION:
Study design This is a single-center, prospective, randomized, placebo-controlled, double-blinded trial in patients undergoing open-heart surgery at Richard M. Ross Hospital - The Ohio State University Medical Center. All study procedures will be done in accordance with institutional and ORRP-IRB guidelines.

Study participants Adult patients undergoing open-heart surgery at Richard M. Ross Hospital - The Ohio State University Medical Center with an American Society of Anesthesiologists (ASA) physical status of I to IV who are scheduled to undergo open-heart surgery at Richard M. Ross Hospital - The Ohio State University Medical Center.

Sample size Eighty-four subjects who give written informed consent to participate in the study and who meet all inclusion and no exclusion criteria will be included in a single treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients aged > 18
* Undergoing primary cardiac surgery requiring sternotomy
* Able to provide a signed written informed consent
* Able to speak, read, and write in English
* American Society of Anesthesiologists (ASA) physical status I-IV

Exclusion Criteria:

* Any documented cognitive or psychological disorders that, in the opinion of the principal investigator, can interfere with the patients' pain perception
* Diabetes Mellitus with documented neuropathic pain
* Vulnerable populations: pregnant females, prisoners, breast feeding
* Contraindication to nerve block: local infections, bleeding disorders, chest wall deformity, allergy to local anesthetic or dexamethasone
* Previous cardiac surgery
* Previous history of chronic pain diseases requiring consistent analgesic therapy for at least 1 month prior to surgery
* Presence of any medical condition that, in the opinion of the principal investigator, should exclude the patient from the study
* BMI ≥ 40 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
OPIOID consumption at 24 hours | 24 hours after block procedure
  To compare the effect of bilateral PIFB on perioperative opioid consumption (MME) during the first 24 hours after surgery between groups
OPIOID consumption during surgery | Surgery length
  To compare the amount of opioid consumption oral MME consumption during surgery between groups
NRS pain score at 48 hours | Up to 48 hours after block procedure
  To compare the NRS (0-10) pain score up to 48 hours
Worst pain score at 48 hours | Up to 48 hours after block procedure
  To compare the worst pain experienced during up to 48-hours after surgery between groups
Incidence nausea and/or vomiting after surgery | Up to 48 hours after block procedure
  To compare the incidence of nausea and/or vomiting up to 48-hours after surgery between both groups
Self-reported satisfaction score at 48 hours | 48 hours after block procedure
  To compare self-reported patient satisfaction up to 48 hours after surgery between both groups
pain-DETECT scores at 90 days | Up to 90 days after block procedure
  To compare the "pain-DETECT" questionnaire scores prior to surgery (baseline) and 30 ± 7, 60 ± 7 and 90 ± 7 days after surgery between groups

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
We estimate that a calculated sample size of 42 patients per group: PN ropivacaine and PN saline (control group)is required for a statistical power of 0.90 and a type I error of 0.05, to detect a 15% reduction (65 μg vs 55 μg, SD=13) in MME use between groups, accounting for 90% successful block rate and 10% of loss to follow-up; a total of 84 patients will be included. The primary outcome of mean MME of pain will be compared between the groups using a two-sample t-test or non-parametric equivalent. Continuous secondary outcomes will be analyzed using the same methods. Categorical secondary outcomes will be analyzed using Chi-square test/Fisher's Exact tests.